CLINICAL TRIAL: NCT02350205
Title: SASS 2 : Self Assembled Skin Substitute for the Autologous Treatment of Severe Burn Wounds in Acute Stage of Burn Trauma.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Veronique Moulin, Researcher, CHU de Quebec-Universite Laval
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOEX 014
Record Dates: First submitted 2015-01-15; First posted 2015-01-29 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Burns
Keywords: Burn wounds; Burns; Skin substitute
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (SASS) (Experimental): Phase A: All patients will receive both Self assembled skin substitute (SASS) and Split-thickness autograft (paired samples sites A+ B). // Phase B: All patients will receive Self assembled skin subsitute (SASS)
  Interventions: Biological: Self assembled skin substitute (SASS)

INTERVENTIONS:
Biological: Self assembled skin substitute (SASS) — All patients in Phase B will receive Self assembled skin substitute (SASS)

SUMMARY:
This clinical trial is designed to assess the safety, effectiveness and benefits of Self Assembled Skin Substitute SASS grafts as a permanent skin replacement for the treatment of full-thickness burn wounds that require permanent coverage where the availability of donor sites is limited.

ELIGIBILITY:
Inclusion Criteria:

* Deep second degree burns or third degree burns over 50% TBSA (Total body surface area) at time of recruitment or as determined by the surgeon;
* Limited availability of donor sites for autografts;
* Consent obtained by the participant or by the appropriate representative in case of inapt prospective participants or minors.

Exclusion Criteria:

* Skin grafting needed only on the face, hands, feet, ears or genital area;
* Connective tissue diseases;
* Hypersensitivity to bovine proteins;
* Coagulation disorders prior being burned;
* Immunodeficiency prior being burned;
* Uncontrolled diabetes prior being burned;
* Permanent wound coverage before SASS grafts are ready;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of graft take site A vs site B (Phase A 17 patients) | < 1 month
  Clinical assessment; Image analysis
Percentage of graft take of all SASS (Phase A+B) | < 1 month
  Clinical assessment
Percentage of graft take according to sites (Phase A+B) | < 1 month
  Clinical assessment

SECONDARY OUTCOMES:
Scar evaluation site A vs site B (Phase A 17 patients) | 3, 6, 12, 24 and 36 months
  Vancouver Scar Scales; Cutometer; Mexameter; Dermascan; Images;
Scar evaluation according to sites (Phase A+B) | 3, 6, 12, 24 and 36 months
  Cutometer; Mexameter; Dermascan; Images;
Incidence of adverse events site A vs site B (Phase A 17 patients) | 24 to 36 months
  Clinical assessment: Infection, Hematoma below the graft, corrective surgery, inclusion of cysts, granulation buds, other
Incidence of adverse events of all SASS (Phase A+B) | 24 to 36 months
  Clinical assessment: Infection, Hematoma below the graft, corrective surgery, inclusion of cysts, granulation buds, other
Quality of life survey (Phase A+B) | 3, 6, 12, 24 and 36 months
  Survey BSHS-B ( brief version of the Burn Specific Health Scale)
Ratio harvested surface vs covered surface (Phase A+B) | 1 month
  Planimetric analysis; Clinical assessment; Images; Image analysis;

CONTACTS AND LOCATIONS:
Overall Officials: Veronique J Moulin, PhD, Principal Investigator — CHU de Quebec
Locations (7):
- Canada (7):
  - Foothill Medcial Centre, Calgary, Alberta
  - Mackenzie Health Science's Centre, Edmonton, Alberta
  - BC Children's Hospital Plastic Surgery Clinic, Vancouver, British Columbia
  - Winnipeg Health Science Center, Winnipeg, Manitoba
  - Hospital for Sick Children (Sickkids), Toronto, Ontario
  - Hôpital Sainte Justine, Montreal, Quebec
  - CHU de Québec - Unité des grands brûlés, Québec, Quebec